CLINICAL TRIAL: NCT02574624
Title: Vitreous Surgery With Intraocular Assistance (VISIA)
Brief Title: Vitreous Surgery With Intraocular Assistance
Acronym: VISIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in finding patients with complex retinal pathology to enroll in this study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Peter A Campochiaro, MD, Professor of Ophthalmology and Neuroscience, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VISIA
Record Dates: First submitted 2015-09-24; First posted 2015-10-14 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Traction Retinal Detachments; Rhegmatogenous Retinal Detachments; Dislocated Intraocular Lens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraocular Assistance (Experimental): Intraocular assistance in patients undergoing standard of care vitreous surgeries
  Interventions: Procedure: Intraocular assistance

INTERVENTIONS:
Procedure: Intraocular assistance — Intraocular assistance with help of surgical assistants during vitreous surgery (VISIA) in patients who require vitreous surgeries as part of standard of care procedure for conditions like retinal detachments, dislocated intraocular lens and glaucoma patients requiring endophotocoagulation.

SUMMARY:
To Assess the Safety of Vitreous surgery with intraocular assistance (VISIA) & to identify and document with video evidence and surgeon's case report forms intraocular maneuvers that are facilitated by VISIA.

DETAILED DESCRIPTION:
Standard care surgery will be done with a few novel additions to facilitate the surgical procedure. Currently 3 ports are inserted by creating holes in the sclera (white part of the eye) to enter into the posterior part of the eye. When complex dissection is needed, a fourth port will be inserted. The assistant will insert light source through the 4th port. This eliminates the need for the surgeon to hold the light in one hand. Hence allows freeing of both hands for the surgeon to use a forceps in one hand to grasp and elevate membranes and a scissors in the other to cut connections between the retina and the membranes. When membranes are particularly thick, it can be difficult to dissect with a single forceps holding up the membrane. In this situation, a 5th port will be inserted allowing the assistant to insert a light source through one and a forceps though another. The surgeon will have a forceps in one hand and a scissors in another making dissection process more efficient.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria to be eligible for study entry:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age ≥18 years
* Subject will have complex retinal pathology for which it is judged that surgical objectives could be facilitated by VISIA

Exclusion Criteria:

Subjects who meet any of the following criteria will be ineligible for study entry:

• Patients with disease processes such as macular pucker and macular hole that are generally well-managed by standard two-handed vitrectomy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is recording of adverse events directly related to VISIA and adverse events unrelated to VISIA. | 4 months

SECONDARY OUTCOMES:
Surgeon's assessment of the benefits and risks of VISIA recorded on the surgical case report form. | 4 months
Assistant's assessment of the benefits and risks of VISIA recorded on the surgical case report form. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No